CLINICAL TRIAL: NCT06339762
Title: ''Invitation to Self-Compassion: Reshaping the Burden of Care in the Light of Self-Compassion Training Given to Relatives of Patients in Palliative Care.''
Brief Title: Self-Compassion Training Given to Relatives of Patients in Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/03-19
Record Dates: First submitted 2024-02-23; First posted 2024-04-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Self-Compassion Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Self-Compassion Training
  Interventions: Behavioral: Self-Compassion Training
- Control (No Intervention): Self-Compassion Training no

INTERVENTIONS:
Behavioral: Self-Compassion Training — Self-Compassion Training
  Arms: Experimental

SUMMARY:
The concept of self-compassion is a concept that has been frequently the subject of research lately and has gained importance along with positive psychology. It is also referred to as self-understanding and self-compassion in the literature. The concept of self-compassion used in our study represents the concept of self-compassion in its original form as used in foreign sources. Compassion is classified according to the source to which it is directed or received. It is suggested that there are three different flows: the feeling of compassion that the individual directs from himself to others, the feeling of compassion he receives from others, and the feeling of compassion that he directs directly to his own self. It means showing oneself the same compassion and understanding one does to others, accepting and being open to one's own pain, and being accepting of oneself without being judgmental. Individuals with self-compassion believe that the difficulties, flaws and shortcomings they experience are normal. At the same time, they are aware that being human has characteristics and that everyone can experience these situations. Individuals may be less compassionate towards themselves than they are towards others. Individuals with self-compassion are as understanding, forgiving and loving towards themselves as they are towards other people.

ELIGIBILITY:
Inclusion Criteria:

* Being an inpatient in the Palliative unit of Erzurum City Center City Hospital
* Not having attended self-compassion training before
* The patient's relatives do not have any obstacle to communication
* Participants who gave informed consent to participate in the study.

Exclusion Criteria:

* Relatives of patients who do not agree to participate in the research,
* The participant must have attended self-compassion training before,
* People have a condition that prevents communication
* The occurrence of a physical or psychological problem in people during the research process
* Patient's relatives want to leave before completing the training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Self-Compassion Scale: | 4 week
  Self-compassion is the individual's ability to show the same compassion to himself as he does to others. The scale, whose original name was "self-compassion scale", was developed by Neff (2003b). The purpose of the scale is to measure individuals' self-compassion levels, that is, their self-compassion levels. The scale consists of 26 items and the questions are evaluated on a 5-point Likert scale. The scale has 6 sub-dimensions: self-compassion, self-judgment, common human experiences, conscious awareness, isolation and over-identification. Cronbach's alpha values of the subscales vary between .78 and .81, and the Cronbach's alpha value of the entire scale is .92.
Care Burden Scale: | 4 week
  It was developed by Zarit, Reever and Bach-Peterson in 1980. In studies, the internal consistency coefficient of the scale was found to be between 0.87 and 0.94, and the test-retest reliability was found to be 0.71 (Zarit, 1990). Turkish validity and reliability study was conducted by İnci and Erdem (2008), and the Cronbach alpha reliability coefficient was found to be 0.95. It is a scale used to evaluate the stress experienced by caregivers of individuals or elderly people in need of care.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No